CLINICAL TRIAL: NCT02790905
Title: Validating the Patient Health Questionnaire-9 (PHQ-9) and Refugee Health Screener-15(RHS-15) Questionnaires to Screen for Depression in Pregnant and Post-partum Migrant Women on the Thai-Myanmar Border
Brief Title: Validating the Patient Health Questionnaire in Pregnant and Post-partum Migrant Women
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1503
Record Dates: First submitted 2016-05-19; First posted 2016-06-06 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: pregnant and post-partum women; Validation questionnaires; Thai-Myanmar border
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to validate the Patient Health Questionnaire-9 (PHQ-9) and the Refugee Health Screener-15 (RHS-15) screening tools for depression in pregnant and post-partum migrant women on the Thai-Myanmar border.

DETAILED DESCRIPTION:
Background: Mental illness affects a significant proportion of women during and after pregnancy. The most common form of mental illness is depression, which can manifest with symptoms such as sadness, loss of pleasure in activities, poor sleep, changes in appetite and, in severe cases, suicide. Depression during or after pregnancy can have profound effects on the mother, her family and wider society. Left untreated, depression can become chronic and recurrent and lead to reduced ability to work and provide care. Children of depressed mothers are at increased risk of poor growth, increased infections and delayed cognitive, behavioural and emotional development. Recognising maternal depression at an early stage and offering effective treatment such as counselling or anti-depressant medication is vital to helping women and minimising impacts on their families. To effectively diagnose depression, a variety of screening tools is available. However, psychometric properties vary across populations and contexts, and tools must be validated locally prior to use. This validation study will be based at the Shoklo Malaria Research Unit (SMRU), which has provided health services and conducted research in rural and disadvantaged populations living on the Thai-Myanmar border for nearly three decades.

Research design: The study will be an observational, cross-sectional validation study. Women will be asked to complete two questionnaires and an interview.

Study population: The study population will be women who are pregnant and post-partum (up to 12 months) attending SMRU antenatal and postnatal clinics at Wang Pha, Mawker Tai and Maela.

Method and technique (survey, interview, observation): The questionnaires will be translated into Burmese and Karen, and back-translated into English to ensure that semantics have been maintained. Pregnant and post-partum women attending antenatal clinics (ANC) and postnatal clinics (PNC) who volunteer to participate will be asked to provide consent. Participants will first be asked to complete two questionnaires: the PHQ-9 and RHS-15. These will be administered by a member of SMRU staff in Karen or Burmese. Participants will then be asked to attend a diagnostic interview conducted by the principal investigator with an interpreter. The principal investigator will be blinded to the results of the PHQ-9 and RHS-15 until completion of the interview.

Anticipated outcomes: The outcomes of this validation study will be measures of validity, reliability, sensitivity, specificity, positive predictive value and negative predictive value for each of the screening tools (PHQ-9 and RHS-15).

Potential value and significance: If the questionnaires are found to be valid in the local population they can be used as a routine screen for depression for all women attending antenatal and postnatal clinics at SMRU. Helping to identify women with depression will enable earlier treatment and minimise the impact of depression on her and her family.

ELIGIBILITY:
Inclusion Criteria:

* Women who are pregnant (at any stage of pregnancy) and post-partum (up to 12 months post-partum)
* Willing and able to give informed consent for participation in the study
* Aged 18 years or over

Exclusion Criteria:

* Deemed by study staff to be acutely unwell and unable to participate
* Known mental illness and undergoing treatment/therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who are pregnant (at any stage of pregnancy) and post-partum up to 12 months post-partum, aged 18 years or over, who are willing and able to participate.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Validity of Patient Health Questionnaire-9 (PHQ-9) | at enrollment
Validity of Refugee Health Screener-15 (RHS-15) questionnaire | at enrollment

SECONDARY OUTCOMES:
Reliability of Patient Health Questionnaire-9 (PHQ-9) | at enrollment
Reliability of Refugee Health Screener-15 (RHS-15) questionnaire | at enrollment
Sensitivity of Patient Health Questionnaire-9 (PHQ-9) | at enrollment
Sensitivity of Refugee Health Screener-15 (RHS-15) questionnaire | at enrollment
Specificity of Patient Health Questionnaire-9 (PHQ-9) | at enrollment
Specificity of Refugee Health Screener-15 (RHS-15) questionnaire | at enrollment
Positive predictive value for each of Patient Health Questionnaire-9 (PHQ-9) | at enrollment
Positive predictive value for each of Refugee Health Screener-15 (RHS-15) questionnaire | at enrollment
Negative predictive value for each of Patient Health Questionnaire-9 (PHQ-9) | at enrollment
Negative predictive value for each of Refugee Health Screener-15 (RHS-15) questionnaire | at enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Fellmeth G, Plugge EH, Carrara V, Fazel M, Oo MM, Phichitphadungtham Y, Pimanpanarak M, Wai NK, Mu O, Charunwatthana P, Nosten F, Fitzpatrick R, Mcgready R. Migrant perinatal depression study: a prospective cohort study of perinatal depression on the Thai-Myanmar border. BMJ Open. 2018 Jan 5;8(1):e017129. doi: 10.1136/bmjopen-2017-017129. PMID 29306876